CLINICAL TRIAL: NCT06155994
Title: Phase I/IIa Study to Evaluate the Safety, Tolerability, Whole-body Distribution, and Preliminary Diagnostic Performance of a Novel 68Ga-labelled Minigastrin Analogue in Patients With Advanced Neuroendocrine Tumours
Brief Title: 68Ga-DOTA-MGS5 PET/CT in Patients With Advanced Neuroendocrine Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT No.: 2020-003932-26
Record Dates: First submitted 2023-11-07; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-10

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group A and B (Experimental): Group A: six patients with advanced medullary thyroid carcinoma
  Group B: six patients with advanced gastroenteropancreatic and bronchopulmonary neuroendocrine tumours
  Interventions: Drug: 68Ga-DOTA-MGS5

INTERVENTIONS:
Drug: 68Ga-DOTA-MGS5 — intravenous administration
  Other Names: 68Ga-labelled minigastrin analogue

SUMMARY:
68Ga-labelled [DOTA0,DGlu1,desGlu2-6,(N-Me)Nle11,1-Nal13]minigastrin (68Ga-DOTA-MGS5) is a novel radiopharmaceutical for intravenous administration for evaluation of the cholecystokinin receptor (CCK2R) status in patients with CCK2R-related malignancies. CCK2R is expressed at high incidence in medullary thyroid carcinomas (92%) and frequently expressed also in gastroenteropancreatic neuroendocrine tumours (GEP-NET, 22%). In this phase I/IIa study the safety of administration and the biodistribution of 68Ga-DOTA-MGS5 will be evaluated in patients with advanced MTC as well as gastroenteropancreatic and bronchopulmonary NET. In addition, the visualization of tumour lesions as well as the absorbed organ and tumour radiation dose will be evaluated. The new positron emission tomography (PET) imaging modality has the potential to improve the diagnostic accuracy in patients with advanced MTC as well as gastroenteropancreatic and bronchopulmonary NET. After successful application in diagnostic imaging, CCK2R targeting with therapeutic radionuclides bears high potential also to improve the therapeutic management of patients with advanced disease.

DETAILED DESCRIPTION:
This is a monocentric, open-label, single dose diagnostic Phase I/IIa study. Due to the very limited number of patients and the rare nature of the disease the study was designed as a combination of phases I and IIa. The main objectives of such an early phase clinical trial are safety and tolerability, pharmacokinetics and - in the case of radiopharmaceuticals - dosimetry aspects. All patients will undergo a diagnostic PET/CT imaging study with 68Ga-DOTA-MGS5. The study population will be divided in two groups:

Group A: In this group six patients with advanced MTC will be injected with a single dose of 68Ga-DOTA-MGS5 to evaluate the safety and tolerability of the intravenous injection as well as the preliminary tumour targeting properties of 68Ga-DOTA-MGS5 in MTC patients. Lesions with focal 68Ga-DOTA-MGS5 uptake not explained by physiologic CCK2R expression will be interpreted as metastatic disease.

Group B: In this group additional six patients with other advanced gastroenteropancreatic and bronchopulmonary NET will be included. Besides confirming the safety and tolerability of the intravenous injection of 68Ga-DOTA-MGS5, the preliminary tumour targeting properties will be characterized also for advanced NET. Again, lesions with focal 68Ga-DOTA-MGS5 uptake not explained by physiologic CCK2R expression will be interpreted as metastatic disease.

In the first six patients (independently of the group) 5-6 PET/CT whole-body examinations at different time points after injection will be acquired to evaluate the whole-body distribution and determine the absorbed organ and tumour radiation doses. From this data set the optimal time window for PET/CT imaging will be established to reduce the number of scans to 2 examinations in the last six patients.

The dosimetry data will allow to identify potential critical organs also for possible therapeutic applications. In addition, for pharmacokinetic characterization, serial venous whole blood samples will be collected in the first six patients after each PET examination and urine samples will be collected.

The screening examinations will be performed up to 16 days prior the imaging study. Only subjects fulfilling all the inclusion and none of the exclusion criteria will be accepted in the study.

The administration of 68Ga-DOTA-MGS5 will be performed using a venous access. 68Ga-DOTA-MGS5 PET/CT imaging at 2-6 time points will be performed using 3D PET/CT.

In the first six patients (independently of the group) additional blood sampling for pharmacokinetic assessments will be performed using a venous access at the opposite arm of the patient and urine collection will be carried out.

If needed, patients may be hospitalised for the study procedures. Such a planned hospitalisation for study purposes will not be considered a SAE.

A first follow-up visit will be performed after the last imaging time point or on the next day after 68Ga-DOTA-MGS5 administration.

A second follow-up safety visit is scheduled at day 7 to 16 after 68Ga-DOTA-MGS5 administration.

The clinical trial ends when the last patient has completed the planned last visit according to protocol.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years, men and women
* Understanding and provision of signed and dated written informed consent by the patient or legally acceptable representative prior to any study-specific procedures
* Karnofsky performance status >70
* Histopathologically diagnosed locally advanced or metastatic MTC with calcitonin level >100 pg/mL after total thyroidectomy or other histologically diagnosed advanced gastroenteropancreatic and bronchopulmonary NET with known metastases
* Patients with an advanced stage of the disease as documented by local or distant metastasis in an alternative imaging procedure such as 68Ga-SSTR-PET/CT or 18F-DOPA-PET/CT, including a contrast enhanced CT performed up to six months before study inclusion
* Male subjects must-agree to use condoms throughout the study period and for 1 month after study termination if their partner is of childbearing potential and is using no contraception. They agree not to donate semen during study period and for 1 month after study termination.
* Women of childbearing potential (WOCBP) must have a negative urine/serum pregnancy test. WOCBP who are sexually active, agree to use highly-effective means of contraception during the study and for at least 6 months post-study treatment. Allowed are accepted and effective non-hormonal methods of contraception and sexual abstinence or vasectomised partners (>3 months previously). Vasectomy has to be confirmed by two negative semen analyses.

Exclusion Criteria:

* Other known co-existing malignancies except patients with a history of malignant tumours in complete remission >3 years, with no evidence of recurrence <5 years
* Participation in any other investigational trial within 3 months of study entry
* Treatment with tyrosine kinase inhibitors within 1 month before study entry
* Organ allograft requiring immunosuppressive therapy
* Renal insufficiency with an eGFR <30 mL/min/1.72m2
* Higher than grade 2 hematotoxicity (CTC >2)
* Clinically abnormal ECG (signs of ischemia, high grade ventricular arrhythmia, high grade supra-ventricular arrhythmia)
* Pregnancy, breast-feeding
* Patients with concurrent illnesses or severe infectious diseases that might preclude study completion
* Patients with bladder outflow obstruction or unmanageable urinary incontinence
* Known hypersensitivity to gallium-68 or to any of the excipients of DOTA-MGS5
* Any condition that precludes raised arms position for prolonged imaging purposes
* Prior administration of a radiopharmaceutical within a period corresponding to 8 half-lives of the radionuclide used on such radiopharmaceutical
* Clinically significant illness or clinically relevant trauma within 3 weeks before the administration of the investigational product
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical safety and tolerability | day -16 to 0 before administration, day 0 to 1 after administration; day 7 to16 after administration
  The assessment of standard safety and tolerability will include physical examination, measurement of vital signes, electrocardiogram, laboratory tests (haematology, blood chemistry, coagulation parameters, semiquantitative urine analysis, pregnancy test in women of childbearing potential, tumour markers). Clinical relevant changes will be reported. Any serious adverse reactions (SAR) and any suspected unexpected serious adverse reaction (SUSAR) related to the study drug defined by the CTCAE v5.0 will be monitored. The tolerability and safety of the administration of a diagnostic dose of 68Ga-DOTA-MGS5 in patients is determined by the absence of increased number of SAR and SUSAR compared to other peptide-based radiotracers.
Whole-body distribution and dosimetry | day 0
  Up to 6 whole-body PET/CT scans will be acquired in the first six patients. The number of scans will be reduced to 2 in the last six patients. PET/CT scans will be used for semiquantitative evaluation of tissues and organs with physiologic tracer uptake by measuring the intensity of tracer uptake with the maximum and mean standardised uptake value (SUVmax, SUVmean). From these measurements time activity curves will be generated and residence times of 68Ga-DOTA-MGS5 in normal organs and tumour lesions, as well as absorbed tumour-to-organ doses and effective whole-body dose will be calculated.
Assessment of pharmacokinetics | day 0
  Venous blood sampling and urine collection for pharmacokinetic assessments will be performed in the first six patients to calculate the half-life of 68Ga-DOTA-MGS5 in blood and quantify the urinary excretion.

SECONDARY OUTCOMES:
Preliminary targeting properties | day 0
  In the PET/CT scans, lesions with focal 68Ga-DOTA-MGS5 uptake not explained by physiologic CCK2R expression will be interpreted as metastatic disease. Lesions that are visually considered as suggestive or malignant are analysed with respect to their SUVmax and SUVmean. The observed tumour lesions will be described (number of lesions, uptake per lesion) and compared with known tumour lesions.
Comparison with other standard imaging modalities | day 0
  The targeting properties of 68Ga-DOTA-MGS5 PET/CT will be compared with other standard imaging modalities such as 18F-DOPA-PET/CT and 68Ga-SSTR-PET/CT (number of lesions, uptake per lesion).
Description of lesion agreement | day 0
  Description of the overall, positive and negative agreement on a lesion-by-lesion basis as well as on a patient basis of 68Ga-DOTA-MGS5 PET/CT relative to the standard imaging procedures overall and for each tumour type.

OTHER OUTCOMES:
HPLC radiochromatography of blood and urine | day 0
  Blood and urine collected for pharmacokinetic assessement will be subjected to HPLC radiochromatography analysis to explore the in vivo stability of 68Ga-DOTA-MGS5. The presence of intact 68Ga-DOTA-MGS5 in blood and urine will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Virgolini, MD, Principal Investigator — Medical University of Innsbruck
Locations (1):
- Department of Nuclear Medicine, Medical University of Innsbruck, Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] von Guggenberg E, di Santo G, Uprimny C, Bayerschmidt S, Warwitz B, Hormann AA, Zavvar TS, Rangger C, Decristoforo C, Sviridenko A, Nilica B, Santo G, Virgolini IJ. Safety, Biodistribution, and Radiation Dosimetry of the 68Ga-Labeled Minigastrin Analog DOTA-MGS5 in Patients with Advanced Medullary Thyroid Cancer and Other Neuroendocrine Tumors. J Nucl Med. 2025 Feb 3;66(2):257-263. doi: 10.2967/jnumed.124.268877. PMID 39819687